CLINICAL TRIAL: NCT00607828
Title: Feasibility of Hypofractionated Stereotactic Radiotherapy in Patients With Hepatocellular Carcinoma
Brief Title: Stereotactic Radiation Therapy in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0337-07-FB; P30CA036727 (NIH)
Record Dates: First submitted 2008-02-01; First posted 2008-02-06 (Estimated); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated stereotactic radiotherapy (SRT) (Experimental): All patients who have had successful implantation of a liver marker will undergo a 4D CT scan for planning SRT. Following transfer to the treatment planning system, the CT scan may be correlated by imaging fusion with MRI for contouring integrated tumor volume (ITV). The planning target volume (PTV) will be defined as ITV plus individualized margins which are determined by a 4D CT scan. Novalis with 6MV photons will be used for imaging guided SRT. Cohorts of 3-6 patients will receive SRT at daily doses of 8, 10, 12, 14 Gy within 2 weeks. The starting daily dose level will be 10 Gy. The marker will be localized by orthogonal X-ray to ensure reproducibility. A continuous respiratory gating will be accomplished with ExacTrac Adaptive Gating system if the required planning target margin is larger than 1 cm based on the 4D CT data.
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo radiotherapy

SUMMARY:
This is a phase I trial studying the side effects and best dose of stereotactic radiation therapy (SRT) in treating patients with advanced liver cancer. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
This is a phase I trial studying the side effects and best dose of stereotactic radiation therapy (SRT) in treating patients with advanced liver cancer. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Participants must have pathologically confirmed hepatocellular carcinoma with at least one tumor with a maximum diameter of ≤ 8 cm and must have Karnofsky performance status ≥ 60% and a life expectancy of at least 12 weeks.

The primary objective is determining the safety of hypofractionated stereotactic radiotherapy in patients with advanced hepatocellular carcinoma by using toxicity profiles described in the Common Terminology Criteria for Adverse Events (CTCAE) V.3.0. Secondary objectives are determining the maximal tolerable SRT dose, objective tumor response rate, the value of 4-Dimensional Computed Tomography (4DCT) in liver cancer planning, and the value of breath gating in liver cancer stereotactic body radiotherapy (SBRT). After completion of study therapy, participants are followed at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced hepatocellular carcinoma (HCC)
* Measurable disease, defined as ≥ 1 unidimensionally target lesion that can be accurately measured by CT scan or MRI according to RECIST and must have a maximum diameter ≤ 8 cm
* Child-Pugh class A-B cirrhotic status
* Karnofsky performance status 60-100%
* Life expectancy ≥ 12 weeks
* White blood cell count (WBC) ≥ 2,000/μL
* Platelet count ≥ 60,000/mm³
* Hemoglobin ≥ 8.5 g/dLINR ≤ 2.3
* More than 6 months since prior myocardial infarction
* Prior systemic chemotherapy allowed
* At least 6 weeks since prior non-radiation local therapy (e.g., surgery, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation)
* Concurrent therapeutic anticoagulation (e.g., warfarin or heparin) allowed provided that no prior evidence of underlying abnormality in Prothrombin time (PT/INR) and partial thromboplastin time (PTT) exists

Exclusion Criteria:

* No known central nervous system (CNS) tumors, including metastatic brain disease
* No malignancy within the past 3 years that is distinct in its primary site or histology from HCC, except for carcinoma in situ of the cervix, treated basal cell carcinoma, or superficial bladder tumors (i.e., Ta, Tis, and T1), or any other cancer that has been curatively treated > 3 years prior to study entry
* No renal failure requiring hemodialysis or peritoneal dialysis
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection > grade 2
  * New York Heart Association (NYHA) class II-IV congestive heart failure
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Uncontrolled hypertension
* Condition that could jeopardize the safety of the patient or study compliance
* No history of variceal bleeding where the varices have not been eradicated or decompressed by shunt placement
* No condition that would prevent the patient from undergoing marker implantation
* Not pregnant or nursing/negative pregnancy test
* No substance abuse, medical, psychological, or social condition that may interfere with the patient's participation in the study or evaluation of the study results
* No prior radiotherapy to the liver

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11-16 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Lin, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 Gy x 5: Dose Level 10 Gy x 5
- 12 Gy x 5: Dose Level 12 Gy x 5
- 14 Gy x 5: Dose Level 14 Gy x 5
Period: Overall Study
Arm/Group | 10 Gy x 5 | 12 Gy x 5 | 14 Gy x 5
Started | 3 | 3 | 1
Completed | 3 | 3 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 Gy x 5 | 12 Gy x 5 | 14 Gy x 5 | Total
Number analyzed (Participants) | 3 | 3 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 00 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 3 | 3 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 3 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 1 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Hypofractionated Stereotactic Radiotherapy in Patients With Advanced Hepatocellular Carcinoma
Description: Toxicity as assessed by NCI CTCAE v3.0 (Adverse Events). Due to delayed toxicities attributable to radiotherapy, all toxicities observed within 1 month after SRT will be scored. Dose limiting toxicity (DLT) is defined as any of following toxicities, that is possibly, probably or definitely related to Stereotactic Radiation Therapy (SRT) occurring within 1 month from the start of treatment:
  1. grade 4 or 5 hepatic
  2. grade 4 or 5 gastrointestinal
  3. grade 4 or 5 thrombocytopenia
  4. grade 4 hepatic liver enzyme elevations persisting for ≥ 5 days
  5. any adverse event requiring interruption of therapy by ≥ 2 weeks (14 calendar days).
Time Frame: Up to 1 month after Stereotactic Radiation Therapy (SRT) treatment
Measure: Count of Participants; unit: Participants
Groups:
- 14 Gy x 5: Dose Level 12 Gy x 5
Arm/Group | 10 Gy x 5 | 12 Gy x 5 | 14 Gy x 5
Number analyzed (Participants) | 3 | 3 | 1
Participants
  Experienced at least 1 Toxicity | 0 | 0 | 1
  Experienced No Toxicities | 3 | 3 | 0

2. Secondary Outcome: Response at 1-month Post SRT
Description: Response rate from tumor measurement at 1-month post-SRT
Time Frame: Measured from first day of SRT to 1-month post SRT.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 Gy x 5 | 12 Gy x 5 | 14 Gy x 5
Number analyzed (Participants) | 3 | 3 | 1
Participants
  PR | 3 | 2 | 0
  SD | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Toxicity data was collected up to 3 months post-RT.
Description: toxicity according Common Terminology Criteria for Adverse Events v.3
Arm/Group | 10 Gy x 5 | 12 Gy x 5 | 14 Gy x 5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 Gy x 5 (N=3) | 12 Gy x 5 (N=3) | 14 Gy x 5 (N=1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase (AST) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Elevated AST
Alanine Transaminase (ALT) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) — Elevated ALT
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Elevated Alkaline phosphatase
Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) — Elevated Bilirubin
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) — Low Grade Fever
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-12-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT00607828/Prot_SAP_000.pdf